CLINICAL TRIAL: NCT03271580
Title: Biofilm Modified Macrophage Phenotype and Function in Diabetic Wound Healing
Status: Terminated | Type: Observational
Why Stopped: Insufficient Staff
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Dr. Sashwati Roy, Professor, Indiana University
Other Study IDs: 1808802536
Record Dates: First submitted 2017-06-12; First posted 2017-09-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Wound; Bacterial Infections; Diabetes Mellitus; Infected Ulcer of Skin
Keywords: Wound healing; Diabetes; Inflammatory cells; Macrophage
MeSH Terms: conditions — Wounds and Injuries; Bacterial Infections; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Wound Vac Sponge, Wound Tissue biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients infected ulcers: Diabetic patients with HbA1c<9 with who have wound 4weeks or longer with infection with following interventions:
  1. Finger prick test for HbA1c measurement
  2. Punch biopsy
  3. VAC sponge collection
  4. Ankle brachial index
  Interventions: Diagnostic Test: Finger prick test for HbA1c measurement; Procedure: Punch Biopsy; Other: Vac Sponge Collection; Other: Ankle Brachial Index
- Diabetic patients non infected Ulcers: Diabetic patients with HbA1c<9 who have wound 4 weeks or longer without infection with following interventions:
  1. Finger prick test for HbA1c measurement
  2. Punch biopsy
  3. VAC sponge collection
  4. Ankle brachial index
  Interventions: Diagnostic Test: Finger prick test for HbA1c measurement; Procedure: Punch Biopsy; Other: Vac Sponge Collection; Other: Ankle Brachial Index

INTERVENTIONS:
Diagnostic Test: Finger prick test for HbA1c measurement — HbA1c measurement with finger prick method
Procedure: Punch Biopsy — Wound site will be anaesthetized, by punch biopsy tissue will be collected, wound site will be monitored for bleeding(if bleeding Cautery will be used to stop bleeding).
Other: Vac Sponge Collection — NPWT sponge which is discarded as biological waste, will be collected for wound macrophage isolation
Other: Ankle Brachial Index — Blood pressure test

SUMMARY:
The purpose of this study is to learn more about biofilm and to see how it affects diabetic wounds. A biofilm can occur if a chronic infection causes bacteria to grow in a slime enclosed group. This grouping of bacteria is called a biofilm.

DETAILED DESCRIPTION:
There is one study visit with a 14-week follow-up that will take place during the participants standard of care visit at the Indiana University Health Comprehensive Wound Center (CWC). The following procedures will take place once your appointment has been completed:

* Informed consent will be signed (if not previously signed)
* A hemoglobin A1c drawn will be taken by research personnel, if one has not been done within the last 90 days to check your average blood sugar level.
* An Ankle Brachial Index (ABI) will be obtained if the participant has a leg wound. This is to ensure that participants have adequate blood flow to your wound. This is a non-invasive test which measures blood pressure in both of the participants arms and ankles.
* Demographics (such as your name and address and phone number, age), medical history, current medications, current standard of care labs, and wound data (measurements, cause of the wound, wound culture, assessments, treatments, and duration) will be recorded. The participant's medical record number will also be recorded.
* A photo of the wound site will be taken.
* Wound Vac Collection - The wound vac sponge will be collected (waste by product of the therapy) by the research staff.
* An optional two 3 mm punch tissue biopsies will be obtained from the participant's provider. To perform the biopsy, the area surrounding the wound will first be numbed using a local anesthetic agent that will be injected at the wound site. Then, a pencil-like instrument will be used to remove a small, thin cylinder of tissue. Each biopsy is about the size of this dot. After the tissue is removed, a sterile gauze will be placed on the area to stop any minor bleeding that may occur. The biopsies will be looked at in the laboratory to look at the microorganisms. You will not receive the results of the completed laboratory analysis. (Note: If two biopsies cannot be obtained per your physician's discretion, only one biopsy, debridement tissue (dead tissue that is removed from your wound) or no tissue will be obtained, and/or culture swabs (your wound will be swabbed with something like a Q-tip to collect cells to test for bacteria or other organisms in the wound) will be collected to test for infection.)

During the 14-week follow-up visit, research staff will review the participant's medical chart to determine the final status of the wound. If the participant does not return to the CWC at 14 weeks, the last CWC visit will be documented as the wound check follow-up. This does not require the participant to return for an extra study visit. This information will only be collected from their medical chart if available:

* Final status of the wound (healing, not healing, healed)
* Wound data (measurements), treatments, and any standard of care labs will be obtained
* A photo of your wound from the medical chart will be obtained (if available)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above years old
2. Willing and able to provide informed consent
3. Willing and able to comply with protocol instructions, including biopsies and study visits
4. Diabetics with an open wound
5. Receiving Negative Wound Pressure Therapy (NPWT)

Exclusion Criteria:

1. Inadequate arterial supply, as evidenced by any of the following (for wounds below the knee):

   1. TcOM < 30mmHg
   2. ABI < 0.7
   3. TBI < 0.6
2. Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-eight diabetic subjects with chronic foot ulcer(s) that are receiving Negative Wound Pressure Therapy (NPWT) will be enrolled. Eighteen subjects will be infected and 10 subjects will be non-infected serving as the control for the study. The inclusion and exclusion criteria were carefully selected to enroll diabetic patients who have wound tissue oxygenation adequate to support wound healing.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Biofilm infection | 14 Weeks
  Biofilm Infection using SEM and RT PCR analysis
macrophage phenotyping | 14 Weeks
  Wound macrophage phenotypes using flowcytometry, RTPCR and RNA Seq

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD, Principal Investigator — Indiana University
Locations (5):
- United States (5):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Davis Heart and Lung Institute, Columbus, Ohio
  - The Ohio State University Hospital East, Columbus, Ohio
  - Comprehensive Wound Care Centers, The Ohio State University Hospital, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breen JD, Karchmer AW. Staphylococcus aureus infections in diabetic patients. Infect Dis Clin North Am. 1995 Mar;9(1):11-24. PMID 7769212
- [Background] Davis SC, Martinez L, Kirsner R. The diabetic foot: the importance of biofilms and wound bed preparation. Curr Diab Rep. 2006 Dec;6(6):439-45. doi: 10.1007/s11892-006-0076-x. PMID 17118226
- [Background] James GA, Swogger E, Wolcott R, Pulcini Ed, Secor P, Sestrich J, Costerton JW, Stewart PS. Biofilms in chronic wounds. Wound Repair Regen. 2008 Jan-Feb;16(1):37-44. doi: 10.1111/j.1524-475X.2007.00321.x. Epub 2007 Dec 13. PMID 18086294
- [Background] Hanke ML, Angle A, Kielian T. MyD88-dependent signaling influences fibrosis and alternative macrophage activation during Staphylococcus aureus biofilm infection. PLoS One. 2012;7(8):e42476. doi: 10.1371/journal.pone.0042476. Epub 2012 Aug 3. PMID 22879997
- [Background] Hanke ML, Heim CE, Angle A, Sanderson SD, Kielian T. Targeting macrophage activation for the prevention and treatment of Staphylococcus aureus biofilm infections. J Immunol. 2013 Mar 1;190(5):2159-68. doi: 10.4049/jimmunol.1202348. Epub 2013 Jan 30. PMID 23365077
- [Background] Neut D, Tijdens-Creusen EJ, Bulstra SK, van der Mei HC, Busscher HJ. Biofilms in chronic diabetic foot ulcers--a study of 2 cases. Acta Orthop. 2011 Jun;82(3):383-5. doi: 10.3109/17453674.2011.581265. Epub 2011 May 11. No abstract available. PMID 21561305
- [Background] Zhao G, Usui ML, Lippman SI, James GA, Stewart PS, Fleckman P, Olerud JE. Biofilms and Inflammation in Chronic Wounds. Adv Wound Care (New Rochelle). 2013 Sep;2(7):389-399. doi: 10.1089/wound.2012.0381. PMID 24527355